CLINICAL TRIAL: NCT03253146
Title: The Role and Mechanism of Vimentin in Sepsis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH ZS1080
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2016-05

CONDITIONS: Sepsis
Keywords: Vimentin; sepsis; immune cells; apoptosis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Within 24 h (the first day of study) after ICU admission, blood samples was collected.Blood was centrifuged at 3,000 rpm for 15 minutes. The supernatants were transferred to Eppendorf tubes and stored at -80°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sepsis: Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection.
  Organ dysfunction can be identified as an acute change in total SOFA score ≥2 points consequent to the infection.
  The baseline SOFA score can be assumed to be zero in patients not known to have preexisting organ dysfunction.
  ASOFA score ≥2 reflects an overall mortality risk of approximately 10% in a general hospital population with suspected infection. Even patients presenting with modest dysfunction can deteriorate further, emphasizing the seriousness of this condition and the need for prompt and appropriate intervention, if not already being instituted.
  In lay terms, sepsis is a life-threatening condition that arises when the body's response to an infection injures its own tissues and organs.
  Interventions: Diagnostic Test: VIM detection
- septic shock: Patients with septic shock can be identified with a clinical construct of sepsis with persisting hypotension requiring vasopressors to maintain MAP ≥65 mm Hg and having a serum lactate level >2 mmol/L (18mg/dL) despite adequate volume resuscitation.
  Interventions: Diagnostic Test: VIM detection

INTERVENTIONS:
Diagnostic Test: VIM detection — VIM expression in serum and lymphocytes detection

SUMMARY:
Sepsis is the most common cause of death in the clinical critically ill patients. We have successfully screened the sepsis biomarkers by clinical proteomics approach and found that Vimentin (VIM) played an important role in the occurrence and development of sepsis. However, the exact mechanism is remaining unclear. In this study, the relationship between the changes of peripheral circulation VIM expression and different stages of sepsis development will be further verified in lager clinical trials, as well as the relationship between VIM expression and apoptosis of immune cells (e.g lymphocytes) will also be clarified. This may indicate that the role of VIM in the cell-mediated immunity apoptosis and inflammation-related pathways. Through the implementation of this study, we can clarify the clinical value of VIM and the mechanism of VIM-mediated immune cell apoptosis during the sepsis development from the molecular level, and determine whether the VIM as a new target for sepsis diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

Sepsis 3.0 was adopted to selected participants

Exclusion Criteria:

Participants were excluded if they were younger than 18 years of age; contracted acquired immunodeficiency syndrome; had reduced polymorphonuclear granulocyte counts (<500 μL-1); died within 24 h after admission to the ICU; refused to participate in the study; or declined treatment during the period of observation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Between july 2016 and december 2017, inpatients were included who were in the Department of critical care medicine of the Peking Union Medical College Hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day survival | 28-day
  The survival time of patients more than 28days is defined as survival. The survival time of patients less than 28days is defined as death.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Su L, Pan P, Yan P, Long Y, Zhou X, Wang X, Zhou R, Wen B, Xie L, Liu D. Role of vimentin in modulating immune cell apoptosis and inflammatory responses in sepsis. Sci Rep. 2019 Apr 5;9(1):5747. doi: 10.1038/s41598-019-42287-7. PMID 30952998